CLINICAL TRIAL: NCT04026568
Title: A Single Dose Pharmaco-Diagnostic for Peripheral Nerve Continuity After Trauma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study investigator left Institution
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STUDY00012040
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Nerve Injury
Keywords: Peripheral nerve trauma; laceration; blast injury; mangled limb
MeSH Terms: conditions — Lacerations; Blast Injuries | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single dose 4AP (Experimental): 15mm opaque capsule containing 10mg of 4-AP
  Interventions: Drug: 4-Aminopyridine
- Placebo (Placebo Comparator): Opaque capsule identical looking to the 4AP placebo pill
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: 4-Aminopyridine — Single drug test for nerve continuity
  Other Names: oral dalfampridine
  Arms: Single dose 4AP
Drug: Placebo oral tablet — Placebo arm
  Other Names: Generic placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the role of 4-aminopyridine (4-AP) on the course of recovery after peripheral nerve traction and/or crush injury. The investigational treatment will be used to test the hypothesis that 4-aminopyridine speeds the often slow and unpredictable recovery after peripheral nerve traction and/or crush injuries.

DETAILED DESCRIPTION:
This proposal contains two distinct aims to be investigated in two similar but distinct groups of patients.

Aim 1: To examine the mechanistic effect of 4AP on the return of sensorimotor function and EDX sensitivity in the setting of nerve dysfunction from orthopaedic trauma. This aim tests the hypothesis that oral one-time administration of 4AP provides transient return of function and EDX sensitivity to the traumatically denervated limb in alert patients with known limb injuries not involving the central nervous system.

Aim 2: To examine the mechanistic effect of 4AP on the return of sensorimotor function and EDX sensitivity in the setting of iatrogenic nerve injury after surgical intervention. This aim tests the identical hypothesis as in Aim 1 in a distinct group of patients, whose nerve dysfunction is the result of a clinical intervention, and whose function before that intervention was intact.

Scientific Background and Gaps

Neurological injury in the form of traction or crush to nerves that control muscles and sensory function is common. Because an understanding of these injuries is only now beginning to emerge, research on potential treatments is an important next step. Through experiments performed on animals with the Acorda Therapeutics, Inc. version of the drug (AMPYRA®), 4-aminopyridine (4-AP) has been strikingly effective in ameliorating the effect of a standardized peripheral nerve crush injury. The peripheral nerve injury used in the experiments was a standard model of peripheral nerve injury used to measure recovery in animals and is a model of peripheral nerve traction and crush injury that has been studied for over thirty years. The investigators have found that:

1. 4-AP administration in a single dose given on day three after the injury led to a drastic reduction in the dysfunction afforded by a crush injury just days after the crush itself.
2. 4-AP treatment's effect was short-lived after a single dose and was, in effect, diagnostic of the potential to recover in a nerve that was crushed but not shattered.
3. Severed nerves show no capacity to recover even with 4-AP treatment.
4. The treatment in a daily regimen led to profound, lasting, permanent improvement in the speed of recovery in these animals.

4-AP is used in some of the most fragile of neurologically-ailing patients and is currently a mainline treatment in the setting of multiple sclerosis (1). Multiple sclerosis patients suffer a demyelinating disorder that causes the stripping of the myelin sheath from around neurons in the peripheral and central nervous system. The myelin covering allows for normal conduction of impulses and, without such covering, impulses are small, impaired, impeded, and ineffective. The recognition that crush injuries to nerves do not simply sever the axonal fibers but also demyelinate some population of nerve cells has led to the idea to study the treatment of peripheral nerve traumatic injuries in humans using 4-AP.

Previous Data

4-AP has been studied in humans since the early 1980s, and principles of safe usage are extremely well established. For the purposes of this proposal, the immediate release formulation of 4-AP, sometimes called fampridine will be referred to as IR 4-AP. The proposed version of the drug used in this study is an extended release formulation of 4-AP, called dalfampridine, which was marketed under the trade name AMPYRA, by Acorda Therapeutics. Recently, this extended release formulation has become available as a generic, which will be referred to as generic AMPYRA or dalfampridine. Essentially identical principles apply whether 4-AP is provided in an orally available immediate release formulation (IR 4-AP) or an orally available sustained release formulation (dalfampridine). The safety of 4-AP appears to be determined solely by serum levels.

It has long been recognized that the most significant safety concern regarding 4-AP is an increased frequency in seizures, which occurs in a small percentage of patients if serum levels exceed 100 ng/ml. Therefore, dosages are chosen to maintain serum levels that do not exceed 50-60ng/ml. In this proposal, 5mg of study drug will be administered once every six hours, for a total dosage per day of 20 mg. This total dose, as indicated by multiple previous studies on immediate release 4-AP, has an excellent safety profile even in the fragile population of patients with multiple sclerosis. A sustained release formulation of 4-AP (AMPYRA®) at this same dose is FDA approved for use in the multiple sclerosis population even with a known risk of seizure activity in these patients.

It is important to note that multiple studies on 4-AP also include patients with chronic stroke, chronic spinal cord injury, transverse myelitis, primary lateral sclerosis, Lambert-Eaton myasthenic syndrome, ocular nystagmus, nonarteritic anterior ischemic optic neuropathy, spinal muscular atrophy, chronic Guillain-Barre syndrome, episodic ataxia Type 2, obstructive sleep apnea and spinocerebellar ataxias. Over 45 clinical trials have been conducted in the US alone (as listed on the Clinicaltrials.gov website). There are also 49 primary publications on clinical trials outcomes on 4-AP, which include patients with multiple sclerosis, chronic spinal cord injury, spinocerebellar ataxias and chronic stroke.

The many trials on 4-AP have been conducted using both immediate release 4-AP and sustained release 4-AP. The difference between the immediate release and sustained release formulations are that the sustained release formulation helps to decrease the peaks and troughs in serum levels that can occur with larger doses of immediate release formulations.

The Study Rationale is to evaluate the role of 4-aminopyridine (4AP) on the diagnosis of complete (severed) vs incomplete (non-severed) peripheral nerve injury (PNI). The investigational treatment will be used to test the hypothesis that 4AP allows the identification of incomplete injuries earlier than standard electrodiagnostic (EDX) and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trauma involving two or less limbs where the continuity of a given peripheral nerve or nerves is unclear on presenting physical examination.
* Closed soft tissue envelope obscuring direct observation of the continuity of the affected nerve.
* Cognitive ability to report sensory and motor deficit during examination.
* Able to complete dosing within four days (96 hours) of nerve injury diagnosis.
* Able to provide informed consent
* Eligible for standard of care plan of monitoring vs surgical exploration of the nerve.
* Adults subject aged 18-90
* Known limb trauma which resulted in nerve injury (aim 1) or post-operative/post intervention nerve injury (aim 2).
* Ability to give written informed consent.
* Capable of safely undergoing electrodiagnostic testing (EDX).
* Availability for all testing days and main trial day.

Exclusion Criteria:

* Not able to complete dosing within four days (96 hours) of nerve injury diagnosis
* Distracting injury which prevents adequate examination.
* Plan for surgical exploration of the nerve during the ensuing 48 hours.
* Plan for surgical exploration of the nerve as part of another surgical procedure within 48 hours of evaluation.
* Intoxication during examination or evidence of cognitive deficit that emerges during examination.
* History of multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of hypersensitivity to AMPYRA® or 4-aminopyridine
* Renal impairment based on calculated GFR (GFR<80 mL/min) This laboratory value is measured in all inpatient trauma patients as part of the standard of care.
* History of difficult compliance with timely follow up or plan to seek care at another institution closer to home.
* Patients outside the age range or unable to consent.
* Patients with a known history of a seizure disorder (4AP overdose can, in selected cases, result in limited seizure activity).
* Patients with a concomitant traumatic brain injury.
* Patients unable to communicate return or loss of sensation.
* Patients unable to exhibit motor control on the affected limb at baseline.
* Patients unwilling to complete the study requirements.
* Patients with injuries too extensive to isolate a single nerve(s) for testing.
* Pregnancy, breastfeeding or incarcerated individuals.
* Patients currently taking organic cat-ion transporter 2 (OCT2) inhibitors, eg. Cimetidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Elfar, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- MS Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The results include both subjective and objective measures. Subjective measures will not be hidden from patients given the nature of measurements. Active discussion of objective measures will wait until final follow up at 20 weeks. Patients can use their subjective assessments in their standard-of-care treatment decisions and with their doctors. Investigators will not inform other physicians except at the consent of patients. Objective test results will not be discussed with treating physicians until 20 weeks. If a patient wants further surgical exploration of an injured peripheral nerve based on subjective return of function (or lack) with members of the study team, a patient conference will be arranged with ethicist and DSMB (Data Safety Monitoring Board). The patient's decision in conjunction with the treating surgeon (not on study team to avoid any conflicts) is to be paramount. Unblinding will also be discussed then with the DSMB.

REFERENCES:
- [Background] Robinson LR. Role of neurophysiologic evaluation in diagnosis. J Am Acad Orthop Surg. 2000 May-Jun;8(3):190-9. doi: 10.5435/00124635-200005000-00006. PMID 10874226
- [Background] Robinson LR. Traumatic injury to peripheral nerves. Muscle Nerve. 2000 Jun;23(6):863-73. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-0. PMID 10842261
- [Background] Wilbourn AJ. The electrodiagnostic examination with peripheral nerve injuries. Clin Plast Surg. 2003 Apr;30(2):139-54. doi: 10.1016/s0094-1298(02)00099-8. PMID 12737349
- [Background] Seddon HJ, Medawar PB, Smith H. Rate of regeneration of peripheral nerves in man. J Physiol. 1943 Sep 30;102(2):191-215. doi: 10.1113/jphysiol.1943.sp004027. No abstract available. PMID 16991601
- [Background] SEDDON HJ. Nerve grafting. Ann R Coll Surg Engl. 1963 May;32(5):269-80. No abstract available. PMID 13987582
- [Background] SUNDERLAND S, BRADLEY KC. Denervation atrophy of the distal stump of a severed nerve. J Comp Neurol. 1950 Dec;93(3):401-9. doi: 10.1002/cne.900930304. No abstract available. PMID 14803568
- [Background] SUNDERLAND S. A classification of peripheral nerve injuries producing loss of function. Brain. 1951 Dec;74(4):491-516. doi: 10.1093/brain/74.4.491. No abstract available. PMID 14895767
- [Background] Korompilias AV, Lykissas MG, Kostas-Agnantis IP, Vekris MD, Soucacos PN, Beris AE. Approach to radial nerve palsy caused by humerus shaft fracture: is primary exploration necessary? Injury. 2013 Mar;44(3):323-6. doi: 10.1016/j.injury.2013.01.004. Epub 2013 Jan 23. PMID 23352153
- [Background] Niver GE, Ilyas AM. Management of radial nerve palsy following fractures of the humerus. Orthop Clin North Am. 2013 Jul;44(3):419-24, x. doi: 10.1016/j.ocl.2013.03.012. Epub 2013 Apr 24. PMID 23827843
- [Background] Li Y, Ning G, Wu Q, Wu Q, Li Y, Feng S. Review of literature of radial nerve injuries associated with humeral fractures-an integrated management strategy. PLoS One. 2013 Nov 8;8(11):e78576. doi: 10.1371/journal.pone.0078576. eCollection 2013. PMID 24250799
- [Background] Rocchi M, Tarallo L, Mugnai R, Adani R. Humerus shaft fracture complicated by radial nerve palsy: Is surgical exploration necessary? Musculoskelet Surg. 2016 Dec;100(Suppl 1):53-60. doi: 10.1007/s12306-016-0414-3. Epub 2016 Nov 30. PMID 27900704
- [Background] Han SH, Hong IT, Lee HJ, Lee SJ, Kim U, Kim DW. Primary exploration for radial nerve palsy associated with unstable closed humeral shaft fracture. Ulus Travma Acil Cerrahi Derg. 2017 Sep;23(5):405-409. doi: 10.5505/tjtes.2017.26517. PMID 29052827
- [Background] Chang G, Ilyas AM. Radial Nerve Palsy After Humeral Shaft Fractures: The Case for Early Exploration and a New Classification to Guide Treatment and Prognosis. Hand Clin. 2018 Feb;34(1):105-112. doi: 10.1016/j.hcl.2017.09.011. PMID 29169591
- [Background] Perry JD. Electrodiagnosis in musculo-skeletal disease. Best Pract Res Clin Rheumatol. 2005 Jun;19(3):453-66. doi: 10.1016/j.berh.2005.01.007. PMID 15939369
- [Background] Korte N, Schenk HC, Grothe C, Tipold A, Haastert-Talini K. Evaluation of periodic electrodiagnostic measurements to monitor motor recovery after different peripheral nerve lesions in the rat. Muscle Nerve. 2011 Jul;44(1):63-73. doi: 10.1002/mus.22023. PMID 21674522
- [Background] Capacio BR, Byers CE, Matthews RL, Chang FC. A method for determining 4-aminopyridine in plasma: pharmacokinetics in anaesthetized guinea pigs after intravenous administration. Biomed Chromatogr. 1996 May-Jun;10(3):111-6. doi: 10.1002/(SICI)1099-0801(199605)10:33.0.CO;2-E. PMID 8792860
- [Background] Elfar JC, Yaseen Z, Stern PJ, Kiefhaber TR. Individual finger sensibility in carpal tunnel syndrome. J Hand Surg Am. 2010 Nov;35(11):1807-12. doi: 10.1016/j.jhsa.2010.08.013. PMID 21050964
- [Background] Sahin F, Atalay NS, Akkaya N, Ercidogan O, Basakci B, Kuran B. The correlation of neurophysiological findings with clinical and functional status in patients following traumatic nerve injury. J Hand Surg Eur Vol. 2014 Feb;39(2):199-206. doi: 10.1177/1753193413479507. Epub 2013 Mar 1. PMID 23456925
- [Background] Sims SE, Engel L, Hammert WC, Elfar JC. Hand Sensibility, Strength, and Laxity of High-Level Musicians Compared to Nonmusicians. J Hand Surg Am. 2015 Oct;40(10):1996-2002.e5. doi: 10.1016/j.jhsa.2015.06.009. Epub 2015 Aug 5. PMID 26253604
- [Background] Chimenti PC, McIntyre AW, Childs SM, Hammert WC, Elfar JC. Prospective cohort study of symptom resolution outside of the ulnar nerve distribution following cubital tunnel release. Hand (N Y). 2015 Jun;10(2):177-83. doi: 10.1007/s11552-014-9688-9. PMID 26034427
- [Background] Chimenti PC, McIntyre AW, Childs SM, Hammert WC, Elfar JC. Combined Cubital and Carpal Tunnel Release Results in Symptom Resolution Outside of the Median or Ulnar Nerve Distributions. Open Orthop J. 2016 May 24;10:111-9. doi: 10.2174/1874325001610010111. eCollection 2016. PMID 27347239
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Roberts C. Modelling patterns of agreement for nominal scales. Stat Med. 2008 Mar 15;27(6):810-30. doi: 10.1002/sim.2945. PMID 17634968
- [Background] Kim J, Farahmand M, Dunn C, Davies Z, Frisbee E, Milla C, Wine JJ. Evaporimeter and Bubble-Imaging Measures of Sweat Gland Secretion Rates. PLoS One. 2016 Oct 21;11(10):e0165254. doi: 10.1371/journal.pone.0165254. eCollection 2016. PMID 27768743
- [Background] Kiistala R, Kiistala U, Parkkinen MU, Mustakallio KK. Local sweat stimulation with the skin prick technique. Acta Derm Venereol. 1984;64(5):384-8. PMID 6208715
- [Background] Park SJ, Tamura T. Distribution of evaporation rate on human body surface. Ann Physiol Anthropol. 1992 Nov;11(6):593-609. doi: 10.2114/ahs1983.11.593. PMID 1476561
- [Background] Buchmann SJ, Penzlin AI, Kubasch ML, Illigens BM, Siepmann T. Assessment of sudomotor function. Clin Auton Res. 2019 Feb;29(1):41-53. doi: 10.1007/s10286-018-0530-2. Epub 2018 May 8. PMID 29737432
- [Background] Cardenas DD, Ditunno J, Graziani V, Jackson AB, Lammertse D, Potter P, Sipski M, Cohen R, Blight AR. Phase 2 trial of sustained-release fampridine in chronic spinal cord injury. Spinal Cord. 2007 Feb;45(2):158-68. doi: 10.1038/sj.sc.3101947. Epub 2006 Jun 13. PMID 16773037
- See also: Hand sensibility, strength, and laxity of high-level musicians compared to nonmusicians — https://www.ncbi.nlm.nih.gov/pubmed/26253604

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Dose 4AP | Placebo
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — study terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subject enrolled from Orthopaedic Trauma service for traumatic peripheral nerve injury.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose 4AP | Placebo | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 53 (0) | 53 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Subjective Return of Sensation
Description: Return of lost sensation after nerve injury attributable to circulating 4-AP. Subjective return of sensation in the injured limb or portion of the limb.
  Patients for this trial are not able to sense in portions of their limbs. The measure will be sensation, measured on the binary scale of yes or no (able to feel the extremity versus unable to feel) This is assessed through clinical examination of the injured limb.
Time Frame: During dosing of drug intervention (5 hours) and 2, 6, 9, 12, 15, 20 weeks post injury
Population: Subject enrolled from Orthopaedic Trauma service following traumatic peripheral nerve injury
Measure: Number; unit: participants
Arm/Group | Single Dose 4AP | Placebo
Number analyzed (Participants) | 0 | 1
participants
  Return of sensation prior to administration of study drug-baseline |  | 0
  Return of sensation 1 hour post study drug administration |  | 0
  Return of sensation 2 hours post study drug administration |  | 0
  Return of sensation 3 hours post study drug administration |  | 0
  Return of sensation 4 hours post study drug administration |  | 0
  Return of sensation 5 hours post study drug administration |  | 0
  Return of sensation 2 weeks post injury |  | 0
  Return of sensation 6 weeks post injury |  | 0
  Return of sensation 9 weeks post injury |  | 0
  Return of sensation 12 weeks post injury |  | NA — Subject not evaluated past 9 weeks post injury due to early termination of the study
  Return of sensation 15 weeks post injury |  | NA — Subject not evaluated past 9 weeks post injury due to early termination of the study
  Return of sensation 18 weeks post injury |  | NA — Subject not evaluated past 9 weeks post injury due to early termination of the study
  Return of sensation 20 weeks post injury |  | NA — Subject not evaluated past 9 weeks post injury due to early termination of the study

ADVERSE EVENTS:
Time Frame: Subject adverse events collected during the period of enrollment which is 9 weeks post injury
Description: Due to early termination of the study, no subjects were enrolled in the 4AP study arm and therefore no subjects were at risk
Arm/Group | Single Dose 4AP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of funding and the investigator and IND holder leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04026568/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04026568/ICF_001.pdf